CLINICAL TRIAL: NCT02509234
Title: Trabectedin and Irinotecan in Pediatric Refractory Sarcomas
Brief Title: Trabectedin and Irinotecan for Refractory Pediatric Sarcomas
Acronym: TrIPReSarc
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: TrI.PReSarc V150429
Record Dates: First submitted 2015-07-01; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma; Recurrent Rhabdomyosarcoma
Keywords: pediatric sarcomas; Ewing sarcoma; rhabdomyosarcoma; soft tissue sarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Combined chemotherapy with trabectedin followed by irinotecan — Day 1:
  Trabectedin 1,1 - 1,5 mg/m²/day i.v.
  Day 3-5 and 10-12:
  Irinotecan 30- 90 mg/m²/day p.o. or i.v.

SUMMARY:
The purpose of the study is to evaluate patients with refractory childhood sarcomas, who have been treated with a combination therapy of trabectedin and irinotecan (within compassionate use), to determine, if this is a promising treatment option with acceptable toxicity and if the results warrant a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults (age10 - 40 yoa) with refractory sarcoma, for which there are presently no further treatment options in EURO-Ewing/ EURAMOS/CWS (i.e. ≥ second relapse in ES, resistance to surgery in osteosarcoma, relapsed rhabdomyosarcoma) and have been treated with a combined chemotherapy of trabectedin and irinotecan (described in intervention)
* existing matched control in existing study databases
* have started of treatment within three months of last progress

Key Exclusion Criteria:

* Patients newly diagnosed or in first relapse.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adults (age10 - 40 yoa) with refractory sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Toxicity during therapy | As long as patient is undergoing therapy/ 6 months
  WHO toxicity grading

SECONDARY OUTCOMES:
Quality of life | 12 months
  Assessment of quality of life at the day before starting the next cycle and at months 3, 6, 9 and 12 after start of treatment, using adapted Karnofsky Score.
Assessment of therapeutic effect | 12 months
  Read out after every two cycles (functional imaging, PET-MRT/PET-CT), evaluation according to RECIST.
Assessment of time to treatment failure | 12 months
  Read out after every two cycles (functional imaging, PET-MRT/PET-CT), evaluation according to RECIST.

OTHER OUTCOMES:
Overall survival in comparison to matched controls. | 12 months
  Comparison of overall survival in a matched pair analysis.
Differences in response rate comparing response rate in Ewing Sarcoma to response rate in Soft Tissue Sarcoma | 12 months
  Statistical comparison of response rate according to RECIST in Ewing Sarcoma vs. Soft Tissue Sarcoma
Event free survival in comparison to matched controls. | 12 months
  Comparison of event free survival in a matched pair analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Burdach, Prof., Study Chair — Kinderklinik München Schwabing - Klinik und Poliklinik für Kinder- und Jugendmedizin, Klinikum Schwabing, Städtisches Klinikum München GmbH und Klinikum Rechts der Isar (AöR) der Technischen Universität München